CLINICAL TRIAL: NCT03774225
Title: Effects Of Physiotherapy Intervention In A Motor Training With Virtual Reality On Motor, Cognitive, Balance And Gait Of Patients With Parkinson Disease: A Randomized Clinical Trial
Brief Title: The Influence of Manual and Verbal Guidance for Therapeutic Results in People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pâmela e Amarílis
Record Dates: First submitted 2018-09-05; First posted 2018-12-12 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-07

CONDITIONS: Parkinson Disease
Keywords: Virtual Reality; International Classification of Functioning; Disability and Health; Rehabilitation; Gait; Balance
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities; Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, single-blind, parallel-group, randomised trial
Who Masked: Investigator
Masking Description: The assessments where conducting by a blind examiner (investigator) in different days of the training. The examinator wasn't know which group the participant would be performing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual and verbal guidance (MVG) (Experimental): The MVG Group will be done by experimental group with the manual and verbal guidance of a physiotherapist using four games of X-Box Kinect system®
  Interventions: Other: Virtual Reality with Manual and Verbal Guidance; Other: Virtual Reality with No Manual and Verbal Guidance; Other: Physical Therapy
- No manual and verbal guidance (NMVG) (Experimental): The NMVG Group will be done by experimental group using four games of X-Box Kinect system® in the presence of a physiotherapist that will care about the safety of the participants without interfere in their moviment pattern.
  Interventions: Other: Virtual Reality with Manual and Verbal Guidance; Other: Virtual Reality with No Manual and Verbal Guidance; Other: Physical Therapy
- Physical Therapy (Active Comparator): The Control Group will be trained by conventional Physical Therapy exercises.
  Interventions: Other: Virtual Reality with Manual and Verbal Guidance; Other: Virtual Reality with No Manual and Verbal Guidance; Other: Physical Therapy

INTERVENTIONS:
Other: Virtual Reality with Manual and Verbal Guidance — Participants will perform 4 balance games during 8 sessions with a manually and verbally assisted by a experient physiotherapist.
  Other Names: Experimental Group with Manual and Verbal Guidance (MVG)
Other: Virtual Reality with No Manual and Verbal Guidance — Participants will perform 4 balance games during 8 sessions in the presence of a experient physiotherapist that will ensure patient safety, providing motivational verbal stimuli, and replicating the feedback provided by the game.
  Other Names: Experimental Group with No Manual and Verbal Guidance (NMVG)
Other: Physical Therapy — Patients of the control group will be trained with balance exercises by a experient physiotherapist.
  Other Names: Control Group

SUMMARY:
A prospective, single-blind, parallel-group, randomised trial was conducted in Sao Paulo, Brazil. Thrid eight People with Parkinson's Disease were recruited and randomly allocated in two groups: Experimental Group (EG), that performed the balance and gait training based on games from Microsoft Xbox Kinect System ® (MXKS) supported by manual and verbal guidance (MVG) provided by a PT and a control group (CG) that performed an identical training with no MVG during the training.

DETAILED DESCRIPTION:
It were recruited PPD in the "Brazil Parkinson Association" (BPA), a no-government association of PD care, where the assessments and intervention were performed from December 2017 to June 2018. The PPD were recruited by randomization from the BPA list of active patients and waiting list for PT intervention.

Outcome measures were obtained at up to three time points: before intervention, after 1 week and after 8 weeks of the end of intervention, the last time point was considered as a follow-up assessment. This study is in agreement with CONSORT guidelines for developing randomised trials . Primary measures was the functional balance evaluation by the Balance Evaluation Systems Test (BESTest) and Rapid Turn Test (RT Test), and gait performance assessed in the six-minute walk test and Gait test in 30 seconds. As secondary measures were used: Unified Parkinson's Disease Rate Scale (UPDRS), 5-Step Standing Passing Test (ST-DP5), International Falls Efficiency Scale (FES-I), Brazilian Version of the Freezing Scale March (FOGQ), Parkinson's Disease Quality of Life Questionnaire (PDQ-39), Geriatric Depression Scale (GDS-15).

All patients performed 8 individual training sessions, under the supervision of a physiotherapist, twice a week for four weeks. Each session had 10 minutes of identical global exercises for both groups, consisting of stretching, muscle strengthening and axial mobility exercises, one serie per session. After these initial 10 minutes, both groups performed an additional 40 minutes of balance training using four XBOX games, four per session, under different conditions for MVG and NMVG.

While the Control Group will be trained by conventional Physical Therapy exercises.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosis according to Parkinson's Disease Society Brain Bank of London criteria
* Active treatment with levodopa
* Classification in stages 1, 2 and 3 according to Hoehn and Yahr Classification

Exclusion Criteria:

* Severe cognitive impairment defined as ≤ 20 in Montreal Cognitive Assessment
* Severe respiratory and / or cardiovascular conditions
* Visual and / or auditory deficit that can not be corrected with orthotics;
* Other previously detected orthopedic or neurological diseases, other than Parkinson's Disease, that may interfere with the individual's performance;
* Previous experience with Microsoft XBOX Kinect® games;
* Be in rehab at another location concomitant with study training.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-07-20 (Estimated)

PRIMARY OUTCOMES:
Change in Functional balance and gait with Best Test | 1 week before beginning the training; after 1 week of the end of training; and after 8 weeks of the ending the training (follow up)
  A scale consisting of 36 items, the score having a variation in four levels, 0 being the worst performance and 3 the best, with a total score of 108. This scale evaluates the balance under six different domains: biomechanical changes, stability / verticality limits, anticipatory postural adjustments, postural responses, sensory orientation and gait stability
Change in Gait with 6 minut walk test | 1 week before beginning the training; after 1 week of the end of training; and after 8 weeks of the ending the training (follow up)
  a gait assessment method that measures the maximum distance a person can walk and measures maximal cardiorespiratory functions
Change in Functional balance with Rapid turn test | 1 week before beginning the training; after 1 week of the end of training; and after 8 weeks of the ending the training (follow up)
  Is a mesure of dynamic balance. The subject tested turns in a complete circle (360 degrees) as faster as it could while time to finshed the turn is recorded. The test is done for both sides (right and left).

SECONDARY OUTCOMES:
Specific motor and non-motor aspects of Parkinson's disease with UPDRS scale | 1 week before beginning the training; after 1 week of the end of training; and after 8 weeks of the ending the training (follow up)
  It's a scale composed of four parts: Part I (non-motor aspects of daily life), Part II (motor aspects of daily life), Part III (motor evaluation) and Part IV (motor complications)
Risk of falls with FES-I scale | 1 week before beginning the training; after 1 week of the end of training; and after 8 weeks of the ending the training (follow up)
  presents questions about the concern with the possibility of falling when performing 16 activities, with respective scores from one to four. The total score can range from 16 (no concern) to 64 (extreme worry)
Endurance with 6 minut walk test | 1 week before beginning the training; after 1 week of the end of training; and after 8 weeks of the ending the training (follow up)
  a gait assessment method that measures the maximum distance a person can walk and measures maximal cardiorespiratory functions

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Brazil Parkinson Association, São Paulo
  - Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy, School of Medicine, University of São Paulo, São Paulo